CLINICAL TRIAL: NCT04091815
Title: Impact of Enhanced Recovery (ERAS) Protocol After Laparoscopic Colorectal Surgery Implementation on Clinical Outcomes
Brief Title: Enhanced Recovery After Laparoscopic Colorectal Surgery Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Egle Kontrimaviciute, MD, PhD, Assoc Prof, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19BMT32
Record Dates: First submitted 2019-08-13; First posted 2019-09-17 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Laparoscopic Colorectal Surgery
Keywords: Enhanced recovery; Multimodal analgesia; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I group - general anaesthesia (Active Comparator): General anesthesia, induction with fentanyl, propofol, roqurium. Maintenance - sevoflurane (BIS ranges 40 - 60), opioids (fentanyl and morphine), roqurium. Intraoperative fluid administration - 2000ml sterofundine, 500ml Gelaspan. 75mg intravenous diclofenac sodium on anesthesia induction, 1000mg intravenous acetaminophen at the start of wound closure. Surgical site infiltration, bupivacaine, 0.25%-10 ml, after the last suture.
  Interventions: Other: Type of anaesthesia
- II group - combined - spinal and general anaesthesia (Experimental): Spinal anesthesia: L3-4 interspace, 27G needle, bupivacaine hyperbaric, 16 mg, morphine sulfate 0.1% - 0.1ml.
  General anesthesia, induction with fentanyl, propofol, roqurium. Maintenance - sevoflurane (BIS ranges 40 - 60), roqurium. Intraoperative fluid administration - 2000ml sterofundine, 500ml Gelaspan. 75mg intravenous diclofenac sodium on anesthesia induction, 1000mg intravenous acetaminophen at the start of wound closure. Surgical site infiltration, bupivacaine, 0.25%-10 ml, after the last suture.
  Interventions: Other: Type of anaesthesia

INTERVENTIONS:
Other: Type of anaesthesia — Two different types of anesthesia general vs combined (spinal and general)

SUMMARY:
The study will assess the impact on quality of care after implementation of the ERAS (Enhanced Recovery After Surgery) protocol for laparoscopic colorectal surgery in Vilnius University Hospital Santaros klinikos. The primary goal of this study is to compare efficacy of two different types of anaesthesia - general and combined (spinal and general), efficacy of multimodal analgesia in both groups, need for rescue analgetics, time to bowel movement, time to ambulation. We also aim to study overall patient satisfaction and measure health-related quality of life, from date of randomisation until the date of hospital discharge, 30 days, 3 months and 6 months post-discharge.

DETAILED DESCRIPTION:
Recovery After Surgery (ERAS) protocol is a multimodal perioperative care pathway designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery, now widely accepted in laparoscopic colorectal surgery.

In laparoscopic colorectal surgery, the ERAS protocol involves an accurate interview with the patient in the preoperative phase aimed at smoking and alcohol cessation, the reduction of preoperative fasting with administration of oral carbohydrates before surgery, use of intestinal preparation for selected cases only, the prophylaxis of thromboembolism, a correct antibiotic prophylaxis, the prevention of intraoperative hypothermia and hypotension, prevention of volume overload, preference for minimally invasive surgery, multimodal analgesia with reduced opioid requirements, local anaesthetics for wound infiltration, prevention of postoperative nausea and vomiting, very limited use of the nasogastric tube, early removal of the urinary catheter, multimodal analgesia to minimize opiate consumption, early postoperative mobilization and early postoperative feeding, to promote rapid recovery of gastrointestinal functions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* scheduled for laparoscopic colorectal surgery.
* patient informed and having accepted the principle of enhanced recovery after surgery.
* patient written consent will be obtained preoperatively for eligible study participants.

Exclusion Criteria:

Preoperative:

* patients who can not comply with the ERAS protocol because they do not understand the language or has a cognitive disorder.
* patients with a documented allergy to nonsteroidal anti-inflammatory drugs and acetaminophen.
* preoperative renal insufficiency (creatinine clearance less than or equal to 30ml/min) or hemodialysis.
* patients with a history of hepatic impairment.
* chronic pain condition that required daily opioid dependence.

Operative:

* conversion to laparotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | From time to PACU admission until discharge. Every 6 hour for first 24-hour, then every 12 hour until 72 hours.
  Number of patients with unsatisfactory pain relief evaluated with visual analogic scale (VAS > 4, with 0-no pain, 10-worst possible pain)

SECONDARY OUTCOMES:
Total post-operative analgetics consumption | From time to PACU admission until 72 hours postoperatively
  Rescue analgesia will be given according to protocol (ketorolac, narcotics).
Time to bowel movement | From time of PACU admission until the date of first documented bowel mowement, assessed 24 hours postoperatively.
  The times it takes for the first bowel movement after postoperative will be measured.
Time oral intake | From time of PACU admission until the date of first documented liquid oral intake.
  The time it takes to start oral liquid intake postoperatively will be measured.
Time to ambulation | From time of PACU admission until the first documented ambulation, assessed 72 hours postoperatively.
  The time it takes for the patient to ambulate successfully after the surgery will be measured.
Time to urinary catheter removal | From time of PACU admission until the date of urinary catheter removed will be measured.
  The time it takes to urinary catheter removal.
Time to hospital discharge | From the date of randomisation until the date of hospital discharge, or 30 days postoperatively hospital postoperatively will be measured.
  The time it takes the patient to be fully discharged from the hospital will be measured.
Incidence of surgical complications | From date of randomisation until the date of hospital discharge, or 30 days postoperatively hospital postoperatively will be measured.
  The incidence of surgical complications will be documented.
Readmission to the hospital | From the date of randomisation until 30 days postoperatively.
  If a patient will be readmitted to the hospital after being fully discharge, the event will be documented.
Post-operative nausea and vomiting | Nausea/vomiting will be evaluated from time to PACU admission until 72 hours postoperatively.
  Nausea will be evaluated by nausea/vomiting score 0 - 3 (0 - no nausea/vomiting, 3 - nausea/vomiting, >3 times per day).
Post-operative pruritus | From time to PACU admission until 72 hours postoperatively.
  Pruritus will be evaluated with a numerical rating scale (0-no pruritus, 10-worst possible pruritus).
Patient satisfaction | From time to PACU admission until discharge, every 6 hours for the first 24-hour, then every 12 hours until 72 hours.
  Overall patient satisfaction as well as satisfaction related to pain, nausea/vomiting and itching management will be measured.This will be measured with a numerical rating scale (0-being worst possible satisfaction and 10-best satisfaction).
A measure of health status with EQ-5D-5L instrument | From the date of randomization until the date of hospital discharge. Then after 30 days, 3 months and 6 months post-discharge.
  The descriptive system to assess a patient's health-related quality of life which comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ instrument VAS scale records the respondent's self-rated health on a vertical, 0-100 visual analog scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Jurate Sipylaite, MD, PhD, Study Chair — Vilnius University, Faculty of Medicine
Locations (1):
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No